CLINICAL TRIAL: NCT03345979
Title: A Phase 3b, Multicenter, Randomized, Double-blind Study to Evaluate the Efficacy and Safety of Aripiprazole Lauroxil or Paliperidone Palmitate for the Treatment of Schizophrenia in Subjects Hospitalized for Acute Exacerbation
Brief Title: A Study of Aripiprazole Lauroxil or Paliperidone Palmitate for the Treatment of Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK9072-A306
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Schizophrenia
Keywords: Alkermes; schizophrenia; aripiprazole lauroxil; ARISTADA; ARISTADA INITIO
MeSH Terms: conditions — Schizophrenia | interventions — aripiprazole lauroxil; Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Treatment Group 1 (Experimental): Regular injections
  Interventions: Combination Product: Aripiprazole Lauroxil
- Treatment Group 2 (Active Comparator): Regular injections
  Interventions: Drug: Paliperidone Palmitate

INTERVENTIONS:
Combination Product: Aripiprazole Lauroxil — Intramuscular injection; study drug provided using a pre-filled syringe
  Other Names: ARISTADA; ARISTADA INITIO
  Arms: Treatment Group 1
Drug: Paliperidone Palmitate — Intramuscular injection
  Other Names: Invega Sustenna
  Arms: Treatment Group 2

SUMMARY:
This study will evaluate the efficacy of initiating treatment of schizophrenia with ARISTADA INITIO plus 30 mg oral aripiprazole followed by a 2-month dose of AL.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of schizophrenia
* Requires acute treatment for symptoms of schizophrenia
* Willing and able to be confined to an inpatient study unit for up to 3-4 weeks
* Has experienced at least one previous hospitalization for schizophrenia
* Has been able to achieve outpatient status for more than 3 months in the past year
* Has a body mass index (BMI) between 18.0 and 40.0 kg/m^2
* Resides in a stable living situation when not hospitalized
* Has an identified reliable caregiver (for example, family member)
* Additional criteria may apply

Exclusion Criteria:

* Poses a current suicide risk
* Pregnant, planning to become pregnant, or breastfeeding
* Initiated first antipsychotic treatment within the past 12 months
* Has received a long-acting injectable antipsychotic in the past 3 months
* Has participated in a clinical study involving any investigational product within the past 3 months, or is currently participating in a clinical study involving an investigational product.
* A positive urine drug test for drugs of abuse
* Additional criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Pathak, MD, Study Director — Alkermes, Inc.
Locations (16):
- United States (16):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Rogers, Arkansas
  - Alkermes Investigational Site, Cerritos, California
  - Alkermes Investigational Site, Culver City, California
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, Lemon Grove, California
  - Alkermes Investigational Site, Hialeah, Florida
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Hoffman Estates, Illinois
  - Alkermes Investigational Site, Flowood, Mississippi
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Las Vegas, Nevada
  - Alkermes Investigational Site, Berlin, New Jersey
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, Garland, Texas
  - Alkermes Investigational Site, Richardson, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sommi RW, Saklad SR, Weiden PJ, Still D, Wang M, Yagoda S. Initiating Aripiprazole Lauroxil: Post Hoc Analysis of Safety and Tolerability of 1-Day and 21-Day Regimens. J Clin Psychiatry. 2024 Aug 12;85(3):23m15132. doi: 10.4088/JCP.23m15132. PMID 39145678
- [Derived] Citrome L, Yagoda S, Bidollari I, Wang M. Safety and Tolerability of Starting Aripiprazole Lauroxil With Aripiprazole Lauroxil NanoCrystal Dispersion in 1 Day Followed by Aripiprazole Lauroxil Every 2 Months Using Paliperidone Palmitate Monthly as an Active Control in Patients With Schizophrenia: A Post Hoc Analysis of a Randomized Controlled Trial. J Clin Psychiatry. 2024 Feb 28;85(1):23m15095. doi: 10.4088/JCP.23m15095. PMID 38416865
- [Derived] Nasrallah HA, Weiden PJ, Walling DP, Du Y, Yao B, Yagoda S, Claxton A. Aripiprazole lauroxil 2-month formulation with 1-day initiation in patients hospitalized for an acute exacerbation of schizophrenia: exploratory efficacy and patient-reported outcomes in the randomized controlled ALPINE study. BMC Psychiatry. 2021 Oct 8;21(1):492. doi: 10.1186/s12888-021-03420-x. PMID 34625041
- [Derived] Weiden PJ, Claxton A, Kunovac J, Walling DP, Du Y, Yao B, Yagoda S, Bidollari I, Keane E, Cash E. Efficacy and Safety of a 2-Month Formulation of Aripiprazole Lauroxil With 1-Day Initiation in Patients Hospitalized for Acute Schizophrenia Transitioned to Outpatient Care: Phase 3, Randomized, Double-Blind, Active-Control ALPINE Study. J Clin Psychiatry. 2020 May 19;81(3):19m13207. doi: 10.4088/JCP.19m13207. PMID 32433835

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 200 patients enrolled and randomized to treatment, there were 195 patients included in the full analysis set. These were patients who randomized, received 1 dose study drug and had at least one post-baseline Positive and Negative Syndrome Scale (PANSS) assessment.
Groups:
- Aripiprazole Lauroxil: Aripiprazole lauroxil (AL)1-day initiation regimen (30mg oral aripiprazole + intramuscular injection aripiprazole lauroxil nano-cyrstalline milled dispersion [AL-NCD]) on day 1, followed by 1064mg intramuscular injection aripiprazole lauroxil on day 8 and every 2 months thereafter
- Paliperidone Palmitate: Paliperidone palmitate (PP) initiation dosing (234mg intramuscular injection on day 1 + 156mg intramuscular injection on day 8), followed by 156mg intramuscular injection paliperidone palmitate every month thereafter
Period: Overall Study
Arm/Group | Aripiprazole Lauroxil | Paliperidone Palmitate
Started | 99 | 101
Completed | 56 | 43
Not Completed | 43 | 58
Not completed — Withdrawal by Subject | 20 | 31
Not completed — Adverse Event | 10 | 11
Not completed — Lost to Follow-up | 8 | 9
Not completed — Lack of Efficacy | 4 | 2
Not completed — Protocol Violation | 1 | 3
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole Lauroxil | Paliperidone Palmitate | Total
Number analyzed (Participants) | 99 | 101 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (9.67) | 43.4 (10.83) | 43.4 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 73 | 76 | 149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 19
  Not Hispanic or Latino | 91 | 90 | 181
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 72 | 78 | 150
  White | 25 | 17 | 42
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Positive and Negative Syndrome Scale (PANSS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Syndrome Scale (PANSS) contains 30 questions, each containing an answer range of 1-7. A total PANSS score can range from between 30 to 210; a higher score indicates a worse disease condition. Population: FAS population includes those who were randomized and received at least one dose of study drug and have at least one post-baseline Positive and Negative Syndrome Scale (PANSS) assessment
  units on a scale
    number analyzed (Participants) | 96 | 99 | 195
    (all) | 94.1 (9.04) | 94.6 (8.41) | 94.4 (8.71)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score at Week 4
Description: Change within treatment groups of Positive and Negative Syndrome Scale (PANSS) total score between baseline and week 4 based on the observed data without imputation for missing data. The PANSS scale contains 30 questions, each containing an answer range of 1-7. A total PANSS score can range from between 30 to 210; a higher score indicates a worse disease condition.
Time Frame: Baseline and 4 weeks
Population: The analysis is based on the subjects who had both baseline and observed week 4 Positive and Negative Syndrome Scale (PANSS) data (160 participants).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Lauroxil | Paliperidone Palmitate
Number analyzed (Participants) | 80 | 80
units on a scale | -17.4 (11.57) | -20.1 (13.72)
Statistical Analysis 1: Comparison: Aripiprazole Lauroxil; Test type: Superiority; p < .001, t-test, 2 sided
Statistical Analysis 2: Comparison: Paliperidone Palmitate; Test type: Superiority; p < .001, t-test, 2 sided

2. Secondary Outcome: Least Squares Mean Change in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 4
Description: Least squares mean change in Positive and Negative Syndrome Scale (PANSS) between at 4 weeks from Mixed Models Repeated Measures (MMRM). The PANSS scale contains 30 questions, each containing an answer range of 1-7. A total PANSS score can range from between 30 to 210; a higher score indicates a worse disease condition
Time Frame: Baseline and 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole Lauroxil | Paliperidone Palmitate
Number analyzed (Participants) | 80 | 80
units on a scale | -17.3 (1.28) | -19.3 (1.25)

3. Secondary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 9
Description: Change within treatment groups from baseline Positive and Negative Syndrome Scale (PANSS) and 9 weeks based on the observed data without imputation for missing data. The PANSS scale contains 30 questions, each containing an answer range of 1-7. A total PANSS score can range from between 30 to 210; a higher score indicates a worse disease condition.
Time Frame: Baseline and 9 weeks
Population: The analysis is based on the subjects who had both baseline and observed week 9 Positive and Negative Syndrome Scale (PANSS) data (131 participants).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Lauroxil | Paliperidone Palmitate
Number analyzed (Participants) | 69 | 62
units on a scale | -19.8 (11.61) | -22.5 (13.98)

4. Secondary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 25
Description: Change within treatment groups at baseline Positive and Negative Syndrome Scale (PANSS) and at 25 weeks based on the observed data without imputation for missing data. The PANSS scale contains 30 questions, each containing an answer range of 1-7. A total PANSS score can range from between 30 to 210; a higher score indicates a worse disease condition
Time Frame: Baseline and 25 weeks
Population: The analysis is based on the subjects who had both baseline and observed week 25 Positive and Negative Syndrome Scale (PANSS) data (99 participants).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Lauroxil | Paliperidone Palmitate
Number analyzed (Participants) | 56 | 43
units on a scale | -23.3 (11.25) | -21.7 (14.37)

5. Secondary Outcome: Least Squares Mean Change in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 9
Description: Least squares mean change from baseline Positive and Negative Syndrome Scale (PANSS) and 9 weeks from Mixed Models Repeated Measures (MMRM).The PANSS scale contains 30 questions, each containing an answer range of 1-7. A total PANSS score can range from between 30 to 210; a higher score indicates a worse disease condition
Time Frame: Baseline and 9 weeks
Population: The analysis is based on the subjects who had both baseline and observed week 9 PANSS data (131 participants).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole Lauroxil | Paliperidone Palmitate
Number analyzed (Participants) | 69 | 62
units on a scale | -18.8 (1.33) | -21.5 (1.34)

6. Secondary Outcome: Least Squares Mean Change in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 25
Description: Least squares mean change in Positive and Negative Syndrome Scale (PANSS) total score at week 25 from Mixed Models Repeated Measures. The PANSS scale contains 30 questions, each containing an answer range of 1-7. A total PANSS score can range from between 30 to 210; a higher score indicates a worse disease condition
Time Frame: Baseline and 25 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole Lauroxil | Paliperidone Palmitate
Number analyzed (Participants) | 56 | 43
units on a scale | -22.0 (1.42) | -21.1 (1.53)

7. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events (AEs)
Time Frame: Up to 25 weeks
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole Lauroxil | Paliperidone Palmitate
Number analyzed (Participants) | 99 | 101
Participants | 69 | 72

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 25 weeks.
Description: Adverse event collection was based on investigator's observation and reporting from subjects.
Arm/Group | Aripiprazole Lauroxil | Paliperidone Palmitate
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/101
Serious Adverse Events (participants affected / at risk) | 8/99 | 7/101
Other Adverse Events (participants affected / at risk) | 39/99 | 50/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole Lauroxil (N=99) | Paliperidone Palmitate (N=101)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 5 (5) | 2 (2)
Psychotic disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (3)
Psychotic symptom (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole Lauroxil (N=99) | Paliperidone Palmitate (N=101)
Injection Site Pain (General disorders) | 17 (28) | 25 (40)
Weight increased (Investigations) | 9 (9) | 17 (17)
Akathisia (Nervous system disorders) | 9 (9) | 11 (13)
Headache (Nervous system disorders) | 8 (9) | 8 (8)
Somnolence (Nervous system disorders) | 4 (4) | 7 (8)
Dystonia (Nervous system disorders) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.

DOCUMENTS (2):
  • Study Protocol (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT03345979/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT03345979/SAP_001.pdf